CLINICAL TRIAL: NCT06879418
Title: Dose Related Effects of Radial Extracorporeal Shock Wave Therapy on Upper Trapezius Trigger Points in Patients With Cervicogenic Headache: A Randomized Controlled Trial
Brief Title: Dose Related Effects of Radial Extracorporeal Shock Wave Therapy on Upper Trapezius Trigger Points in Patients With Cervicogenic Headache.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: MTI University (Other)
Responsible Party: Principal Investigator, Radwa Fayek Hammam, Lecturer of Basic Science, Faculty of Physical Therapy, MTI University., MTI University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: P.T.REC/012/005500
Record Dates: First submitted 2025-02-03; First posted 2025-03-17 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2024-10

CONDITIONS: Cervicogenic Headache
Keywords: shock wave therapy
MeSH Terms: conditions — Post-Traumatic Headache | interventions — Extracorporeal Shockwave Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group A (Experimental): Low dose shock wave therapy plus strengthening and stretching exercise.
  Interventions: Other: Low dose shock wave therapy plus strengthening and stretching exercise for upper trapezius
- Group B (Experimental): Medium dose shock wave therapy on upper trapezius trigger points plus strengthening and stretching exercise for upper trapezius
  Interventions: Other: Medium dose shock wave therapy plus strengthening and stretching exercise for upper trapezius
- Group C (Sham Comparator): Sham shock wave therapy plus strengthening and stretching exercises
  Interventions: Other: sham shock wave therapy plus strengthening and stretching exercise for upper trapezius

INTERVENTIONS:
Other: Low dose shock wave therapy plus strengthening and stretching exercise for upper trapezius — Patients will receive 2000 shocks, 1 bar (energy flux density 0.045 mj/mm2) at frequency 10 MHz on upper trapezius trigger points plus strengthening and stretching exercises for upper trapezius.
  Arms: Group A
Other: Medium dose shock wave therapy plus strengthening and stretching exercise for upper trapezius — patients will receive 2000 shock with 4 bars (Energy flux density 0.18 mj/mm2) at frequency 10 MHz on upper trapezius trigger points plus strengthening and stretching for upper trapezius
  Arms: Group B
Other: sham shock wave therapy plus strengthening and stretching exercise for upper trapezius — patients will receive 2000 shock with energy flus density 0.00 on upper trapezius trigger points plus strengthening and stretching exercise for upper trapezius.
  Arms: Group C

SUMMARY:
A randomized double blinded controlled trial will be conducted to determine and compare the effects of low and medium dose radial extracorporeal shock wave therapy on upper trapezius trigger points in patients with cervicogenic headache. Data will be collected at base line and at the end of the treatment program. Participants will be assigned randomly into three groups Group (A) will receive 2000 shock waves at frequency 10 MHz and 0.045 mj/mm2 flux density plus strengthening and stretching exercise for upper trapezius muscle.

Group (B) will receive 2000 shock waves at frequency 10 MHz and 0.18 mj/mm2 energy flux density plus strengthening and stretching exercise for upper trapezius muscle.

Group (C) will receive sham shock wave therapy plus strengthening and stretching exercise for upper trapezius muscle.

ELIGIBILITY:
Inclusion Criteria:

* Symptoms of mechanical neck pain lasting for more than three months
* Skeletal muscle with a palpable taut band
* Hypersensitive point inside the taut band with the ability to reproduce referred pain when the sensitive spot is palpated,
* Joint soreness in at least one of the upper cervical spine's joints (c1-c3)
* Unilateral discomfort that originates in the neck and radiates to the frontotemporal area
* Pain that is made worse by moving the neck
* Headaches that occur at least once a week for a duration longer than three months.

Exclusion Criteria:

* Other primary headaches (i.e., migraine, tension-type headache)
* Bilateral headaches,
* Other defined cervical problem such as fracture, dislocation, skin disease, illness that is inflammatory, neural illness, vertebrobasilar insufficiency, a birth defect, tumor, or infection.

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 135 (Actual)
Dates: Start 2025-03-01 (Actual); Primary Completion 2025-08-30 (Actual); Study Completion 2025-09-15 (Actual)

PRIMARY OUTCOMES:
Henry Ford Hospital Headache disability inventory (HDI) | before the first session and after the last session (Four weeks)
Upper trapezius electromyographic activity | before the first session and after the last session (Four weeks)

CONTACTS AND LOCATIONS:
Locations (1):
- Modern University for Technology and Information, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided